CLINICAL TRIAL: NCT05986058
Title: Preliminary Efficacy of a Technology-based Physical Activity Intervention for Older Korean Adults During the COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Soonhyung Kwon, Doctoral Student, University of Illinois at Urbana-Champaign
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 21916
Record Dates: First submitted 2022-12-14; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Health; Physical Function
Keywords: Physical activity intervention; Older adults

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hybrid PA intervention (Experimental): The PA intervention implemented 1-hour sessions for 12 weeks focusing on improving (1) body muscle, (2) body flexibility, (3) muscle endurance, and (4) body balance. The 12-week hybrid PA intervention was concurrently deployed in-person at a senior center and at-home through a web-based modality.
  Interventions: Behavioral: Golden Circle

INTERVENTIONS:
Behavioral: Golden Circle — The original Golden Circle project was deployed in response to the COVID-19 pandemic and the need to implement remote social services in South Korea. Golden Circle had the aim of building a case management model using a healthcare-oriented automation system based on wearable devices (smartwatches and mobile applications). Through innovative system expansions, the goals were to promote healthful CVH and physical function and cultivate self-care management skills in older Korean adults.

SUMMARY:
This study tested preliminary efficacy of a hybrid (web-based and center-based) PA intervention combining use of a smartwatch and mobile application. The 12-week hybrid PA intervention included 120 older Korean adults and was concurrently implemented in-person at the local senior center and at-home through a web-based modality. Overall, increases were evident in systolic/diastolic blood pressure, total cholesterol, and high-density-lipoprotein at posttest, with decreases seen for triglyceride levels. Participants showed improvements in muscular function and cardiopulmonary endurance.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 and over
* enrolled member at the participating senior center for at least three years
* fluent in Korean

Exclusion Criteria:

* younger than 60 years old
* less than three years enrollment at the senior center
* cannot read and speak Korean

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Cardiovascular health | Pre (baseline) and posttest (through study completion, 12 weeks later from the baseline)
  systolic and diastolic blood pressure, total cholesterol, high-density lipoprotein, and triglycerides

SECONDARY OUTCOMES:
Physical function | Pre (baseline) and posttest (through study completion, 12 weeks later from the baseline)
  muscular function and cardiopulmonary endurance

CONTACTS AND LOCATIONS:
Locations (1):
- Mokdong Senior Welfare Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
It requires the data agreement from the director (Noh-Suk Park).